CLINICAL TRIAL: NCT05082714
Title: Tocilizumab Versus Baricitinib in Hospitalized Patients With Severe COVID-19: an Open-label, Randomized Controlled Trial
Brief Title: Tocilizumab Versus Baricitinib in Patients With Severe COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Argyris Tzouvelekis, Associate Professor of Respiratory Medicine, Head Department of Respiratory Medicine, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATTKPATRASCOVID19
Record Dates: First submitted 2021-10-18; First posted 2021-10-19 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: COVID-19
Keywords: COVID-19; Acute Respiratory Distress Syndrome; PaO2/FiO2; Tocilizumab; Baricitinib
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome | interventions — tocilizumab; baricitinib

STUDY DESIGN:
Intervention Model Description: Non-inferiority trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tocilizumab (Experimental): tocilizumab plus usual care
  Interventions: Drug: Tocilizumab
- baricitinib (Experimental): baricitinib plus usual care
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Tocilizumab — tocilizumab 8mg/kg single infusion (a second infusion within 48 hours can be applied upon clinician's discretion)
  Arms: tocilizumab
Drug: Baricitinib — The baricitinib intervention consists of baricitinib at a dose of 4 mg/day (given daily for up to 14 days or until discharge from hospital, whichever occurred first); however, 2 mg/day will be given if the patient has a baseline eGFR of 30 to less than 60 mL/min/1·73 m2
  Arms: baricitinib

SUMMARY:
The aim of this study is to investigate whether baricitinib is non-inferior to tocilizumab in severe COVID-19.

DETAILED DESCRIPTION:
Patients with COVID-19 will be assigned to one of the two arms on 1:1 ratio based on the time point that PaO2/FiO2<200 will be observed. Patients aged 18 years or older with PaO2/FiO2 <200 at any time during their hospitalization will be included in the analysis irrespective of values in inflammatory markers, such as CRP and ferritin. Exclusion criteria will be: age<18 years, pregnancy, glomerular filtration rate<30 and application of mechanical ventilation prior patients' transfer to our Hospital. Each patient or the patient's legally authorized representative provided written or witnessed oral informed consent.

Day 1 will be considered the first day that PaO2/FiO2<200 will be identified. Treatment with either tocilizumab or baricitinib will start from day 1. Primary and secondary outcomes will be assessed in the days described below.

This study aims to investigate whether baricitinib is non-inferior to tocilizumab in patients with severe COVID-19. Two hundred fifty one (n=251) patients will be enrolled based on the following assumptions: 1) HR θ 1, 2) HR θο 1.5, 3) overall probability of event (primary end point) 0.6 (based on previous records of our hospital), 4) power 80%, 5) type I error α 5%.

ELIGIBILITY:
Inclusion Criteria:

- COVID-19, PaO2/FiO2<200

Exclusion Criteria:

- Age<18 years, Pregnancy, Glomerular filtration rate<30, Application of mechanical ventilation prior patients' transfer to our Hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2022-06-04 (Actual)

PRIMARY OUTCOMES:
Mechanical ventilation or death by day 28 | day 28

SECONDARY OUTCOMES:
Time to discharge over the 28-day period | day 28
World Health Organization scale at day 10 [range from 0 (not infected) to 10 (dead)] | day 10

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Patras, Department of Respiratory Medicine, Pátrai, Greece

IPD SHARING:
Plan to Share IPD: Yes
data will be available upon request